CLINICAL TRIAL: NCT01389934
Title: Infusion of a Local Anaesthetic in the Surgical After Modified Radical Mastectomy With Expander
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Lourdes Ferreira, Osakidetza/Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MASTEC-002
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2011-07

CONDITIONS: Local Anesthetic
Keywords: levo-bupicaine; Radical; Mastectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Women of this group be infused saline 2 ml / h for 48h.
  Interventions: Drug: Placebo
- levo-bupicaine (Experimental): Women of this group will be infused L-bupivacaine 0.50% 2 ml / h for 48h.
  Interventions: Drug: levo-bupicaine

INTERVENTIONS:
Drug: levo-bupicaine — Women of this group will be infused L-bupivacaine 0.50% 2 ml / h for 48h after intervention
  Arms: levo-bupicaine
Drug: Placebo — Women of this group be infused saline 2 ml / h for 48h.
  Arms: Control

SUMMARY:
Background: The use of local anesthetics as a supplement to conventional techniques in breast surgery is widely reported in the literature. Currently there is controversy regarding the efficacy of surgery for breast infusion of local anesthetic after surgery. The aim of this study demonstrate the efficacy of administering a local anesthetic into the surgical bed of women operated radical mastectomy for breast cancer for the control of postoperative pain.

Material and methods: double-blind randomized clinical trial. The investigators recruited patients who underwent modified radical mastectomy that met inclusion and exclusion criteria. The intervention group were infused with L-bupivacaine 0.50% 2 ml/h for 48 hours, and saline control group at 2 ml/h during surgery and anesthetic technique 48 hours. Local anesthetic and rescue medication was identical in both groups.

Statistical analysis: The baseline patient characteristics of the patients were analyzed by Chi square or Student t always meet criteria of normality, otherwise it will use the Mann-Whitney. To determine the effectiveness of treatment as well as pain scale adverse events will be held on chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with operable breast cancer, which will be submitted to modified radical mastectomy
* Sign informed consent.

Exclusion Criteria:

1. Mastectomy without lymphadenectomy
2. Over 80 years
3. Cognitive impairment and patients with serious psychiatric disorders before diagnosis of the cancer process
4. Severe liver or kidney disease
5. Patients allergic or intolerant to any of the drugs used in the study protocol.
6. Regular users of analgesics or narcotics

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
effectiveness of administering levo-bupicaine to control postoperative pain. | 48 hours
  the control postoperative pain will be measured by a a patient satisfaction scale (very good, good, fair, bad, very bad)

SECONDARY OUTCOMES:
Decreased consumption of other analgesics | 48 hours
  We will measure the number of rescue doses of each drug (acetoaminphen, metamizol, dexketoprofen and morphine) We will include all minor adverse effects (nausea, vomiting ...) as severe (sedacion..) and their resolution.

CONTACTS AND LOCATIONS:
Locations (1):
- Txagorritxu Hospital, Vitoria-Gasteiz, Alava, Spain

REFERENCES:
- [Derived] Ferreira Laso L, Lopez Picado A, Antonanzas Villar F, Lamata de la Orden L, Ceballos Garcia M, Ibanez Lopez C, Pipaon Ruilope L, Lamata Hernandez F, Valero Martinez C, Aizpuru F, Hernandez Chaves R. Cost-effectiveness analysis of levobupivacaine 0.5 %, a local anesthetic, infusion in the surgical wound after modified radical mastectomy. Clin Drug Investig. 2015 Sep;35(9):575-82. doi: 10.1007/s40261-015-0316-4. PMID 26305021
- [Derived] Ferreira Laso L, Lopez-Picado A, Lamata L, Ceballos Garcia M, Ibanez Lopez C, Pipaon Ruilope L, Lamata Hernandez F, Antonanzas Villar F, Valero Martinez C, Aizpuru F, Hernanz Chaves R. Postoperative analgesia by infusion of local anesthetic into the surgical wound after modified radical mastectomy: a randomized clinical trial. Plast Reconstr Surg. 2014 Dec;134(6):862e-870e. doi: 10.1097/PRS.0000000000000762. PMID 25415108